CLINICAL TRIAL: NCT02275091
Title: Identifying Children With Diabetes Type 1 at High Risk for Cardiovascular Disease.
Brief Title: Children With Diabetes at Risk for Heart Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Collaborators: Howard University (Other)
Responsible Party: Principal Investigator, Evgenia Gourgari, M.D., Assistant Professor of Pediatric Endocrinology, Georgetown University
Other Study IDs: 2014-0755
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Complications
Keywords: Children; Cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples will be collected through study completion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes: Children with diabetes type 1 , 12-21 years old
- Healthy: Healthy children 12-21 years old

SUMMARY:
Patients with type 1 diabetes type 1 (DM1) have increased risk of death due to heart disease and stroke. These cardiovascular conditions (CVD) are the leading cause of death in patients with DM1 younger than 40 years of age and up to 35% of all persons with DM1 will die before age 55 from CVD. Strategies are needed to help identify adolescents with DM1 at risk for CVD so that interventions to prevent heart disease and stroke can be undertaken.

DETAILED DESCRIPTION:
Patients with type 1 diabetes and healthy controls will have evaluation of their lipid profile. Arterial stiffness, heart rate variability and adiposity measurements will be done in patients with type 1 diabetes and healthy controls. Blood pressure and heart rate will be recorded. 50 ml of urine will be collected from patients and controls.

All studies will be performed as a single outpatient visit at Georgetown University.

ELIGIBILITY:
Inclusion Criteria:

Diabetes type 1 or Healthy

Exclusion Criteria:

Taking medications that lower cholesterol Duration of type 1 diabetes < 1 year.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with diabetes type 1 and healthy children
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
small LDL particles | This is an observational cross sectional study. Samples will be collected through study completion, on average of 6 years duration.
  Blood test, based on NMR

CONTACTS AND LOCATIONS:
Overall Officials: Evgenia Gourgari, Principal Investigator — Georgetown University
Locations (1):
- Georgetown-Howard Universities Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Gourgari E, Ma J, Playford MP, Mehta NN, Goldman R, Remaley AT, Gordon SM. Proteomic alterations of HDL in youth with type 1 diabetes and their associations with glycemic control: a case-control study. Cardiovasc Diabetol. 2019 Mar 28;18(1):43. doi: 10.1186/s12933-019-0846-9. PMID 30922315
- [Derived] Gourgari E, Playford MP, Campia U, Dey AK, Cogen F, Gubb-Weiser S, Mete M, Desale S, Sampson M, Taylor A, Rother KI, Remaley AT, Mehta NN. Low cholesterol efflux capacity and abnormal lipoprotein particles in youth with type 1 diabetes: a case control study. Cardiovasc Diabetol. 2018 Dec 19;17(1):158. doi: 10.1186/s12933-018-0802-0. PMID 30567548